CLINICAL TRIAL: NCT00949455
Title: A Phase II/III, Randomised, Two-Arm, Comparison of Maintenance Lapatinib Versus Placebo After First-Line Chemotherapy in Patients With HER1 and/or HER2 Overexpressing Locally Advanced or Metastatic Bladder Cancer [LaMB]
Brief Title: A Double Blind Randomised Study of Lapatinib and Placebo in Metastatic TCC of the Urothelium
Acronym: LaMB
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000640393; OCTG-LaMB; BL-2007-02; EUDRACT-2007-001826-28; EU-20929
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Bladder Cancer
Keywords: stage IV bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral lapatinib ditosylate once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate
- Arm II (Placebo Comparator): Patients receive oral placebo once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally
  Other Names: Tykerb; Tyverb
  Arms: Arm I
Other: Placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether lapatinib ditosylate is more effective than a placebo in killing tumor cells.

PURPOSE: This randomized phase II/III trial is studying how well lapatinib ditosylate works compared to a placebo in treating patients with stage IV bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival in patients with HER1- and/or HER2-overexpressing stage IV bladder cancer who have been randomized to maintenance therapy with lapatinib ditosylate or placebo following first-line chemotherapy.

Secondary

* Compare overall survival between these patient groups.
* Evaluate the safety and tolerability of the regimens in these patients.
* Assess and compare quality of life between these patient groups.

OUTLINE: This is a multicenter study. Patients are stratified according to ECOG performance status and response to first line chemotherapy (complete or partial response vs stable disease). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral lapatinib ditosylate once daily in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo once daily in the absence of disease progression or unacceptable toxicity.

Patients undergo quality of life assessment by EORTC QLQ-C30 at baseline and every 4 weeks during study treatment.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the bladder

  * Stage IV disease
  * Metastatic or locally advanced disease
* HER1- and/or HER2-positive disease, defined by the following criteria:

  * 2+ or 3+ intensity on IHC
* Able to commence the study treatment within 10 weeks of completing chemotherapy
* Must have achieved objective response or stable disease following 4-8 courses of first-line chemotherapy

  * No progression with first-line chemotherapy for metastatic disease
  * Any widely accepted chemotherapy regimen for bladder cancer allowed
  * Patients who did not receive cisplatin are eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* ANC ≥ 1.0 x 10^9/L
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 75 x 10^9/L
* ALT/AST < 2 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Serum creatinine ≤ 3.0 ULN AND/OR creatinine clearance ≥ 30 mL/min
* LVEF ≥ 50% (as assessed by quantitative echocardiogram or MUGA)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No current active hepatic or biliary disease, except for any of the following:

  * Gilbert's syndrome
  * Asymptomatic gallstones
  * Liver metastases
  * Stable chronic liver disease per investigator assessment
* No known hypersensitivity to the study medication
* No history of prior or concurrent other neoplasms, except for:

  * Any non life-threatening tumours that have been curatively treated.
  * Prostate cancer isolated to the prostate gland
* No significant cardiac disease, including any of the following:

  * Angina pectoris
  * Severe cardiac arrhythmia requiring medication
  * Severe conduction abnormalities
  * Clinically significant valvular disease
  * Cardiomegaly
  * Prior myocardial infarction
  * Ventricular hypertrophy
  * Congestive heart failure
  * Poorly uncontrolled hypertension (resting diastolic blood pressure > 115 mm Hg)
  * Other cardiomyopathy
* No serious intercurrent medical or psychiatric illness
* No serious active infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 1 line of prior chemotherapy for metastatic or locally advanced disease (neoadjuvant/adjuvant chemotherapy allowed)
* No more than 10 weeks since first-line chemotherapy
* No prior lapatinib ditosylate
* No prior radiotherapy to the indicator lesion(s) (newly arising lesions in previously irradiated areas allowed)
* At least 14 days since prior and no concurrent CYP3A4 inducers, including but not limited to, any of the following:

  * Antibiotics (all rifamycin class agents [e.g., rifampicin, rifabutin, rifapentine])
  * Anticonvulsants (phenytoin, carbamazepine, barbiturates [e.g., phenobarbital])
  * Oral glucocorticoids (cortisone [> 50 mg], hydrocortisone [> 40 mg], prednisone [> 10 mg], methylprednisolone [> 8 mg], dexamethasone [> 2 mg²])
  * St. John's wort or modafinil
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including but not limited to, any of the following:

  * Antibiotics (clarithromycin, erythromycin, troleandomycin)
  * Antifungals (itraconazole, ketoconazole, fluconazole [>150 mg daily], voriconazole)
  * Antiretrovirals/protease inhibitors (delavirdine, nelfinavir, amprenavir, ritonavir, indinavir, saquinavir, lopinavir)
  * Calcium channel blockers (verapamil, diltiazem)
  * Antidepressants (nefazodone, fluvoxamine)
  * Gastrointestinal agents (cimetidine, aprepitant)
  * Grapefruit, grapefruit juice
* At least 6 months since prior and no concurrent amiodarone
* No concurrent radical or curative therapy (radiotherapy or surgery) at the end of first-line treatment (palliative radiotherapy allowed)
* No other concurrent experimental or investigational drugs
* No other concurrent anticancer treatment, including cytotoxic or specific immune therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2009-03; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Disease Progression - at least 20% increase in the sum of longest diameters of target lesions.

SECONDARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Powles, MD, MRCP, Principal Investigator — Queen Mary University of London
Locations (27):
- United Kingdom (27):
  - Barts and the London NHS Trust, London, England
  - NHS Grampian - Aberdeen Royal Infirmary, Aberdeen
  - Basildon and Thurrock University Hospital NHS Trust - Basildon Hospital, Basildon
  - University Hospitals Birmingham NHS Foundation Trust - Birmingham University Hospital, Birmingham
  - Royal Bournemouth and Christchurch NHS Foundation Trust - Royal Bournemouth Hospital, Bournemouth
  - University Hospitals Bristol NHS Trust - Bristol University Hospital, Bristol
  - Cambridge University Hospitals NHS Trust - Addenbrooke's Hospital, Cambridge
  - Mid Essex NHS Trust - Broomfield Hospital, Chelmsford
  - Colchester University Hospitals NHS Trust, Colchester
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - Derby Hospitals NHS Trust - Royal Derby Hospital, Derby
  - NHS Greater Glasgow and Clyde - The Beatson, Glasgow
  - Calderdale and Huddersfield NHS Trust - Huddersfield Royal Infirmary, Huddersfield
  - Ipswich Hospital NHS Trust, Ipswich
  - University Hospitals of Leicester NHS Trust, Leicester
  - Clatterbridge Centre for Oncology NHS Trust, Liverpool
  - Guys & St Thomas' Hospital NHS Trust - Guys Hospital, London
  - Imperial Healthcare NHS Trust, London
  - Royal Marsden NHS Trust, London
  - South Tees NHS Trust - James Cook University Hospital, Middlesbrough
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle
  - Northampton General Hospitals NHS Trust, Northampton
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sherwood Forest Hospitals NHS Trust - Kings Mill Hospital, Nottingham
  - Portsmouth Hospitals NHS Trust - Queen Alexandra Hospital, Portsmouth
  - Barking, Havering and Redbridge NHS Trust - Queens Hospital, Romford
  - Taunton and Somerset NHS Trust - Musgrove Park Hospital, Taunton

REFERENCES:
- [Derived] Bellmunt J, Werner L, Bamias A, Fay AP, Park RS, Riester M, Selvarajah S, Barletta JA, Berman DM, de Muga S, Salido M, Gallardo E, Rojo F, Guancial EA, Bambury R, Mullane SA, Choueiri TK, Loda M, Stack E, Rosenberg J. HER2 as a target in invasive urothelial carcinoma. Cancer Med. 2015 Jun;4(6):844-52. doi: 10.1002/cam4.432. Epub 2015 Feb 26. PMID 25720673